CLINICAL TRIAL: NCT07407361
Title: Radiographic, Histological and Immunohistochemical Evaluation of Allograft, Xenograft, and Combined Grafting in Maxillary Sinus Floor Augmentation: A Prospective Randomized Clinical Study
Brief Title: Comparison of Allograft, Xenograft and Combined Grafting in Maxillary Sinus Augmentation
Acronym: SINUS-GRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Sefa Colak, Associate Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-KAEK-118
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Posterior Maxillary Atrophy; Maxillary Sinus Augmentation
Keywords: Maxillary sinus augmentation; Bone grafts; Dental implants
MeSH Terms: interventions — Transplantation, Homologous; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Histological and immunohistochemical evaluations were performed by a blinded examiner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Experimental): Patients received dental implant placement without sinus augmentation. Bone biopsy samples were obtained during implant placement for histological and immunohistochemical evaluation.
  Interventions: Procedure: Dental Implant Placement Without Sinus Augmentation
- Allograft Group (Experimental): Patients underwent lateral maxillary sinus augmentation using allograft material prior to dental implant placement. Bone biopsies were obtained at implant placement for histological and immunohistochemical analyses.
  Interventions: Procedure: Lateral Maxillary Sinus Augmentation with Allograft
- Xenograft Group (Experimental): Patients underwent lateral maxillary sinus augmentation using xenograft material prior to dental implant placement. Bone biopsies were obtained at implant placement for histological and immunohistochemical analyses.
  Interventions: Procedure: Lateral Maxillary Sinus Augmentation with Xenograft
- Combined Graft Group (Experimental): Patients underwent lateral maxillary sinus augmentation using a combination of allograft and xenograft materials prior to dental implant placement. Bone biopsies were obtained at implant placement for histological and immunohistochemical analyses.
  Interventions: Procedure: Lateral Maxillary Sinus Augmentation with Combined Graft

INTERVENTIONS:
Procedure: Lateral Maxillary Sinus Augmentation with Allograft — Lateral sinus floor elevation was performed using allograft material prior to dental implant placement.
  Arms: Allograft Group
Procedure: Lateral Maxillary Sinus Augmentation with Xenograft — Lateral sinus floor elevation was performed using xenograft material prior to dental implant placement.
  Arms: Xenograft Group
Procedure: Lateral Maxillary Sinus Augmentation with Combined Graft — Lateral sinus floor elevation was performed using a combination of allograft and xenograft materials prior to dental implant placement.
  Arms: Combined Graft Group
Procedure: Dental Implant Placement Without Sinus Augmentation — Dental implant placement was performed without sinus augmentation. Bone biopsy samples were obtained from the implant site during implant placement for histological and immunohistochemical evaluation.
  Arms: Control Group

SUMMARY:
This prospective randomized clinical study evaluates and compares three different grafting approaches (allograft, xenograft, and combined grafting) used in lateral maxillary sinus augmentation prior to dental implant placement.

Patients with posterior maxillary bone deficiency (residual bone height ≤4 mm) undergoing sinus lift surgery were randomly assigned to one of three grafting groups. Cone-beam computed tomography (CBCT) was used to assess bone height before surgery, immediately after grafting, and at 6 months. During implant placement at 6 months, bone biopsy samples were collected from the grafted sites for histological and immunohistochemical evaluation.

The study aims to assess vertical bone gain, graft height stability, and biological bone healing using osteocalcin, osteopontin, and RUNX2 markers. The results are intended to provide clinically relevant information regarding the volumetric and biological behavior of different graft materials used in maxillary sinus augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Patients presenting with posterior maxillary edentulism requiring dental implant rehabilitation.
* Residual alveolar bone height of 4 mm or less, indicating the need for lateral maxillary sinus augmentation.
* Patients suitable for lateral sinus lift surgery based on clinical and radiographic evaluation.
* Ability to provide written informed consent.

Exclusion Criteria:

* Systemic conditions that could affect bone healing (e.g., uncontrolled diabetes, metabolic bone diseases).
* History of radiotherapy or chemotherapy to the head and neck region.
* Active sinus pathology or chronic sinusitis.
* Heavy smoking (more than 10 cigarettes per day).
* Pregnancy or lactation.
* Use of medications known to affect bone metabolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Vertical Bone Height Gain | 6 months
  Vertical bone height gain following lateral maxillary sinus augmentation, measured using cone-beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Graft Height Loss | 6 months
  Change in grafted bone height between early postoperative and 6-month CBCT measurements.
Histological New Bone Formation | 6 months
  Qualitative and semi-quantitative histological evaluation of new bone formation in bone biopsy samples obtained during implant placement.
Immunohistochemical Expression of Osteogenic Markers | 6 months
  Immunohistochemical expression of osteocalcin, osteopontin, and RUNX2 in bone biopsy samples obtained from grafted sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University Faculty of Dentistry, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.